CLINICAL TRIAL: NCT06816966
Title: Systemic Treatments (Chemotherapy-immunotherapy) Based Split-course Adaptive Hypofractionated Radiotherapy for Extensive-stage SCLC: CISART Study
Brief Title: Chemotherapy-immunotherapy-based Split-course Adaptive Hypofractionated Radiotherapy for Extensive-stage SCLC
Acronym: CISART
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, ChenCheng, Cheng Chen, Fujian Medical University Union Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023YF056-02
Record Dates: First submitted 2025-01-16; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Small-cell Lung Cancer
Keywords: Radiation; split; hypofractionated radiotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy-immunotherapy-based split-course adaptive hypofractionated radiotherapy (Experimental): Each cycle of chemotherapy and immunotherapy is synchronized with a 5 Gy dose of radiotherapy, which is precisely targeted at the gross tumor located within the thoracic cavity. The delineation of the target is adaptively adjusted based on the volumetric reduction of the tumor observed at each treatment session.
  Interventions: Radiation: split-course adaptive hypofractionated radiotherapy

INTERVENTIONS:
Radiation: split-course adaptive hypofractionated radiotherapy — Each treatment cycle comprises a solitary radiotherapy session, which allows for its integration with chemotherapy and immunotherapy. The radiotherapy sessions are scheduled at three-week intervals, thereby affording extended recovery periods for normal tissues. An adaptive radiotherapy plan is implemented for each cycle, enabling precise adjustments to the treatment target area in response to the reduction in tumor volume.

SUMMARY:
This study is a prospective, single-arm, phase Ⅱ trial evaluating the safety and efficacy of Chemotherapy-immunotherapy-based split-course adaptive hypofractionated radiotherapy for extensive-stage SCLC

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) represents the most aggressive and metastatic form of lung carcinoma, particularly in its extensive stage1. SCLC is initially highly chemotherapy sensitive, yet it is paradoxically characterized by nearly ubiquitous metastatic relapse and secondary chemoresistance2. Despite the incorporation of immune checkpoint inhibitors (ICIs) has led to improvements in survival, the benefit is only modest, with an overall survival (OS) improvement of approximately 3-5 months, and the median OS has yet to surpass two years3. This highlights the need for innovative combination strategies. Although consolidative thoracic radiotherapy (TRT) has shown promise in improving local control and two-year survival in ES-SCLC patients with residual intrathoracic disease after first-line chemotherapy 4-6, the efficacy of TRT remains uncertain in the era of immunotherapy. RAPTOR (NCT04402788) is an ongoing phase Ⅱ/Ⅲ trial evaluating the addition of TRT to the usual maintenance therapy with atezolizumab in ES-SCLC patients with a partial response (PR)/stable disease (SD). Given that TRT is administered exclusively to selected patients who have demonstrated a positive response to first-line treatment without disease progression（PD）, a significant proportion of patients are ineligible for TRT due to disease progression. ES-SCLC typically presents with a high tumor burden and bulky thoracic lymph nodes which are the most dominant failure site after chemotherapy or chemoimmunotherapy. According to multiregion sequencing, it is reported that treatment-naive SCLC exhibited clonal homogeneity at distinct tumour sites, whereas a multitude of subclones driven by the most recent common ancestor at clinically overt recurrence, which markedly increases spatial and intratumour heterogeneity7. Considering of initial chemotherapy and radiation sensitivity of SCLC and potential synergistic effects of radiotherapy and immunotherapy, investigator hypothesized that add primary thoracic site RT to first-line chemoimmuntherapy may help killing more clonal tumor cells and enhancing systemic disease control. Whereas it must balance the specific toxicity risks of combined therapy to avoid systemic therapy interruption. Based on the findings of split-course SBRT based on systemic therapy (3S) in for locally advanced rectal cancer（NCT05176964）and borderline resectable pancreatic cancer (NCT04289792) in the institution，this study designed as a single-centre, single- arm, prospective phase Ⅱ trial in subjects with treatment- naïve ES-SCLC to treated with EP regimen chemotherapy, PD-L1/1 inhabitors and split-course hypofractionated radiotherapy (SCHR) as first-line therapy. Patients will be synchronously treated with etoposide/platinum (E/P) doublet plus ICIs and SCHR (4-6 fractions×5 Gy). Chemotherapy and ICIs start on days 1,2,3 and day 8 of every 21-day cycle, respectively. A single dose of 5 Gy radiotherapy may be administered either during a three-day chemotherapy cycle or within a two-day window preceding or following the cycle, taking into account the necessary time for radiotherapy planning and potential scheduling constraints such as weekends.Split-course hypofractionated radiotherapy will be response-adaptively delivered in 4-6 treatments to primary lesion, thoracic lymph nodes in thoracic cavity, adjacent involved supraclavicular and cervical lymph nodes because of shrinkage of bulky tumor. Chemotherapy interval spanning weeks not only allow for greater recovery of normal tissue following an injury from initial bulky-area radiation, but may also maximize potential synergies resulting from concomitant immune-oncology approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Any pathologic confirmation of ES-SCLC at any site, either primary or metastases.
2. Patients must have measurable disease and 3 or fewer observable liver metastases.
3. If there is a pleural effusion, patients will be eligible if thoracentesis is cytologically negative or if pleural fluid is too small a volume to effectively sample by thoracentesis and does not show increased metabolic activity on CT/PET imaging
4. Age greater than or equal to 18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
6. Adequate normal organ and bone marrow function
7. The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
8. Life expectancy greater than six (6) months
9. If the autoimmune disease is not active for over 3 years and the patient is not receiving immunosuppressive treatment such as methotrexate or steroids above a dose equivalent to 10 mg prednisone daily, the patient is eligible.
10. Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible.
11. Patients with controlled type 1 diabetes mellitus on a stable insulin regimen are eligible.
12. Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations are excluded only if they have active disease with acute exacerbation and on immunosuppressive medications within the 12 months prior to enrollment. They are eligible otherwise.
13. Severe, active co-morbidity defined as follows: Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of radiation, chemotherapy and ICIs or that may affect the interpretation of the results or render the patient at high risk from treatment complications;
14. Active tuberculosis;
15. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease.
16. Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.

Exclusion Criteria:

1. Metastatic disease invading the liver (> 3 metastases)
2. Patients with malignant pleural and/or pericardial effusions
3. Prior radiotherapy in the thorax that would result in overlapping RT fields
4. Active autoimmune disease, including, but not limited to: systemic lupus erythematosus; rheumatoid arthritis; inflammatory bowel disease (e.g. Crohn's, ulcerative colitis); vascular thrombosis associated with antiphospholipid syndrome; Wegener's granulomatosis; Sjogren's syndrome; Guillain-Barre syndrome; multiple sclerosis; vasculitis; or glomerulonephritis.
5. Known immunosuppressive disease, for example history of bone marrow transplant or chronic lymphocytic leukemia (CLL);
6. Chronic obstructive pulmonary disease (COPD) requiring chronic oral steroid therapy of > 10 mg prednisone daily or equivalent at the time of registration. Inhaled corticosteroids are not exclusionary;
7. Unstable angina and/or congestive heart failure requiring hospitalization within the last 3 months;
8. History of recent myocardial infarction within 6 months prior to registration.
9. Clinically significant interstitial lung disease;
10. History of allogeneic organ transplant;
11. Patients positive for human immunodeficiency virus (HIV) on effective anti-retroviral therapy with undetectable viral load within 6 months and a stable regimen of highly active anti-retroviral (HAART) HIV-positive patients must have no requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
6-month Progression-Free Survival rate | Time from consent to any documented progression or death due to any cause, whichever occurs first, assessed up to 6 months.
  6-month Progression-Free Survival rate from consent.
Safety | Up to 6 months
  For each patient, the maximum severity reported for both immune mediated and non-immune mediated adverse events will be used in the summaries. Adverse events will be summarized regardless of relationship to protocol treatment as assessed by the investigator. All adverse events, adverse events leading to withdrawal, interruption or modification of protocol treatment, grade >= 3 adverse events, and serious adverse events will be summarized. Deaths and cause of death will be summarized. The rate of treatment-related adverse events using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, version [v.]5.0) will be reported with the frequency and severity (e.g., type, grade, and attribution). All adverse events will be classified by the relationship to treatment.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  Time from consent to any documented death due to any cause.
Failure pattern | Up to 2 years
  Record the first site of recurrence based on this treatment modality.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital,, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Survial and safety Survival data, adverse events and failure patterns.
Supporting Information: Study Protocol, CSR
Time Frame: To be made public in the form of a published article about 1 year after the trial is completed
Access Criteria: Researchers who have approval from an Institutional Review Board (IRB).

REFERENCES:
- [Background] Jeremic B, Shibamoto Y, Nikolic N, Milicic B, Milisavljevic S, Dagovic A, Aleksandrovic J, Radosavljevic-Asic G. Role of radiation therapy in the combined-modality treatment of patients with extensive disease small-cell lung cancer: A randomized study. J Clin Oncol. 1999 Jul;17(7):2092-9. doi: 10.1200/JCO.1999.17.7.2092. PMID 10561263
- [Background] Slotman BJ, van Tinteren H, Praag JO, Knegjens JL, El Sharouni SY, Hatton M, Keijser A, Faivre-Finn C, Senan S. Use of thoracic radiotherapy for extensive stage small-cell lung cancer: a phase 3 randomised controlled trial. Lancet. 2015 Jan 3;385(9962):36-42. doi: 10.1016/S0140-6736(14)61085-0. Epub 2014 Sep 14. PMID 25230595
- [Background] Horn L, Mansfield AS, Szczesna A, Havel L, Krzakowski M, Hochmair MJ, Huemer F, Losonczy G, Johnson ML, Nishio M, Reck M, Mok T, Lam S, Shames DS, Liu J, Ding B, Lopez-Chavez A, Kabbinavar F, Lin W, Sandler A, Liu SV; IMpower133 Study Group. First-Line Atezolizumab plus Chemotherapy in Extensive-Stage Small-Cell Lung Cancer. N Engl J Med. 2018 Dec 6;379(23):2220-2229. doi: 10.1056/NEJMoa1809064. Epub 2018 Sep 25. PMID 30280641
- [Background] Bernabe-Caro R, Chen Y, Dowlati A, Eason P. Current and Emerging Treatment Options for Patients With Relapsed Small-cell Lung Carcinoma: A Systematic Literature Review. Clin Lung Cancer. 2023 May;24(3):185-208. doi: 10.1016/j.cllc.2023.01.012. Epub 2023 Feb 8. PMID 36907793
- [Background] Rudin CM, Brambilla E, Faivre-Finn C, Sage J. Small-cell lung cancer. Nat Rev Dis Primers. 2021 Jan 14;7(1):3. doi: 10.1038/s41572-020-00235-0. PMID 33446664